CLINICAL TRIAL: NCT00564538
Title: A Study Comparing Thymoglobulin to Tacrolimus in Liver Transplant and Impact on Renal Function
Brief Title: A Study of Thymoglobulin and Tacrolimus in Liver Transplant
Acronym: thymo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Nebraska (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 424-07
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Liver Transplantation; Liver Disease; Immunosuppression
Keywords: liver transplant
MeSH Terms: conditions — Liver Diseases | interventions — Antilymphocyte Serum; thymoglobulin; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients in arm 1 will receive induction with thymoglobulin at time of transplant with delayed initiation of tacrolimus
  Interventions: Drug: anti-thymocyte globulin (rabbit)
- 2 (Active Comparator): patients in arm 2 will not receive thymo induction at time of transplant and will have immediate initiation of tacrolimus
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: anti-thymocyte globulin (rabbit) — 1.5mg/kg per dose with the first dose initiated in the operating room prior to reperfusion of the transplanted liver. It will then be administered again on post operative day #1, 3 and 5 for a total cumulative dose of 6mg/kg.
  Other Names: thymoglobulin
  Arms: 1
Drug: tacrolimus — Tacrolimus will be administered orally on post op day #1 as per standard of care.
  Other Names: prograf
  Arms: 2

SUMMARY:
The purpose of this study is to compare kidney function, long term patient and graft survival, and incidence of acute rejection in liver transplant recipients between one group receiving thymoglobulin induction and delayed initiation of tacrolimus and another group of liver transplant recipients having immediate administration of tacrolimus without any induction immunosuppression.

DETAILED DESCRIPTION:
Renal insufficiency following liver transplantation in adult recipients is a major cause of morbidity and a major contributor to mortality. One of the key factors contributing to this renal dysfunction is the use of calcineurin inhibitors. There is some evidence to suggest that the first 7-10 days following liver transplantation are crucial in terms of renal function and the ability to avoid the use of nephrotoxic agents such as calcineurin inhibitors may have a significant impact on long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Primary liver transplant recipient with Model for End Stage Liver Disease (MELD) criteria documentation
* Over 18 years of age
* Signed informed consent form
* if female of childbearing potential: Must not be lactating Must have negative serum pregnancy test on study day 0 Must have agreed on a reliable and acceptable form of contraception during the study
* sexually active males must be practicing an acceptable form of contraception

Exclusion Criteria:

* Multiple organ transplants
* Prior solid organ or bone marrow transplant recipients
* Fulminant hepatic failure
* Status 1 transplants
* Liver transplant candidates with greater than 6 weeks of dialysis
* Patients who in the opinion of the Investigator are not eligible for thymo induction at the time of transplant
* Recipients of investigational therapy within 90 days prior to transplant
* Know contraindication to administration of rabbit anti-thymocyte globulin
* Patients whose medical condition is such that the physician feels it would not be in their best interest to participate in the study
* Patients who are unwilling to have a Glofil nuclear medicine scan at specified time points
* History of malignancy within 5 years with the exception of:
* Adequately treated localized squamous or basal cell carcinoma of the skin without evidence of recurrence, and /or
* Hepatocellular carcinoma

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-12; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of renal function via Glo-Fil nuclear medicine scan and laboratory parameters | Post operative day #1, month 6 and month 12

SECONDARY OUTCOMES:
patient and graft survival, incidence of acute rejection, incidence of active CMV disease, incidence of other infections, any adverse events or serious adverse events associated with the use of thymo induction therapy | post op days 1-6, months 3,6, 9, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Grant, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] 1. Fisher NC, Nightingale PG, Gunson BK, Lipkin GW, JM. N. Chronic renal failure following liver transplantation: a retrospective analysis Transplantation 1998; 66 (1): 59. 2. Gonwa TA, Mai ML, Melton LB, et al. End-stage renal disease (ESRD) after orthotopic lvier transplantation (OLTX) using calcineurin-based immunotherapy. Transplantation 2001; 72: 1934. 3. Moreno JM, Cuervas-Mons V, Rubio E, et al. Chronic renal dysfunction after liver transplantation in adult patients: prevelance, risk factors, and impact on mortality. Transplant Proc 2003; 35 (5): 1907.